CLINICAL TRIAL: NCT01468350
Title: A Double-Blind, Placebo-Controlled, Crossover Study in Subjects With Cerebral Palsy to Evaluate the Safety and Tolerability and the Effect on Sensorimotor Function of Dalfampridine-ER
Brief Title: Safety and Tolerability of Dalfampridine in Subjects With Cerebral Palsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DALF-CP-1002
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Results first posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-05

CONDITIONS: Cerebral Palsy (CP)
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- (PART A) AB: dalfampridine-ER 10mg then placebo (Placebo Comparator): Each subject randomized to the AB arm will receive a single witnessed dose of (A) dalfampridine-ER 10 mg, and a single witnessed dose of (B) placebo, two days apart
  Interventions: Drug: dalfampridine-ER 10mg; Other: Placebo
- (PART A) BA: placebo then dalfampridine-ER 10mg (Placebo Comparator): Each subject randomized to the BA arm will receive a single witnessed dose of (B) placebo, and a single witnessed dose of (A) dalfampridine-ER 10 mg, two days apart
  Interventions: Drug: dalfampridine-ER 10mg; Other: Placebo
- (PART B) AB: dalfampridine-ER 10mg then placebo (Placebo Comparator): Each subject randomized to the AB arm will receive multiple doses of (A) dalfampridine-ER 10mg and multiple doses of (B) placebo
  Interventions: Drug: dalfampridine-ER 10mg; Other: Placebo
- (PART B) BA: Placebo then dalfampridine-ER 10mg (Placebo Comparator): Each subject randomized to the BA arm will receive multiple doses of (B) placebo, and multiple doses of (A) dalfampridine-ER 10mg
  Interventions: Drug: dalfampridine-ER 10mg; Other: Placebo

INTERVENTIONS:
Drug: dalfampridine-ER 10mg
Other: Placebo

SUMMARY:
A double-blind, placebo-controlled, crossover study in subjects with cerebral palsy (CP) to evaluate the safety and tolerability and the effect of dalfampridine extended release (ER) tablets on sensorimotor function

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of CP
* No previous use of any dalfampridine formulation
* Ability to perform all the required study procedures. Subjects should be capable of fully extending and flexing both hands

Exclusion Criteria:

* Presence of any progressive neurological disease
* Severe CP defined as the requirement to use a wheelchair at all times and a care taker for constant assistance in daily activities. This definition includes spastic quadriplegia
* Pregnant or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-12; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Carrazana, MD, Study Director — Acorda Therapeutics
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - UCLA/Orthopaedic Hospital Center for Cerebral Palsy, Los Angeles, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Kennedy Krieger Institute at Johns Hopkins University, Baltimore, Maryland
  - Detroit Clinical Research Center, Farmington Hills, Michigan
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - University of Missouri at Columbia, Columbia, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Bethoux F, Fatemi A, Fowler E, Marciniak C, Mayadev A, Waksman J, Zackowski K, Suarez G, Blight AR, Rabinowicz AL, Carrazana E. Safety, Tolerability, and Sensorimotor Effects of Extended-release Dalfampridine in Adults With Cerebral Palsy: A Pilot Study. Clin Ther. 2017 Feb;39(2):337-346. doi: 10.1016/j.clinthera.2016.12.015. Epub 2017 Jan 25. PMID 28131322

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part A, 11 subjects enrolled and randomized. 6 subjects randomized into Sequence BA (placebo - dalfampridine-ER) and 5 randomized into Sequence AB (dalfampridine-ER - placebo). Part B, 24 subjects enrolled and randomized. 12 subjects randomized into Sequence BA (placebo - dalfampridine-ER) and 12 into Sequence AB (dalfampridine-ER - placebo).
Groups:
- (PART A) Placebo Then Dalfampridine-ER 10mg: Each subject randomized to the BA arm will receive a single witnessed dose of (B) placebo, and a single witnessed dose of (A) dalfampridine-ER 10 mg, two days apart
  Day 1, visit 2, subjects will receive placebo. Day 3, visit 3, subjects will receive dalfampridine-ER 10mg
- (PART A) Dalfampridine-ER 10mg Then Placebo: Each subject randomized to the AB arm will receive a single witnessed dose of (A) dalfampridine-ER 10 mg, and a single witnessed dose of (B) placebo, two days apart
  Day 1, visit 2, subjects will receive dalfampridine-ER 10mg. Day 3, visit 3 subjects will receive placebo
- (PART B) Placebo Then Dalfampridine-ER 10mg: Each subject randomized to the BA arm will receive multiple doses of (B) placebo, and multiple doses of (A) dalfampridine-ER 10mg
  Day 1, visit 2, subjects will be given 15 tablets of placebo taken twice daily for 7 days and an additional 1 tablet for 1 day. Day 15, visit 4, subjects will be given 15 tablets dalfampridine-ER taken twice daily for 7 days and an additional 1 tablet for 1 day
- (PART B) Dalfampridine-ER 10mg Then Placebo: Each subject randomized to the AB arm will receive multiple doses of (A) dalfampridine-ER 10mg and multiple doses of (B) placebo
  Day 1, visit 2, subjects will be given 15 tablets dalfampridine-ER taken twice daily for 7 days and an additional 1 dose for 1 day. Day 15, visit 4, subjects will be given 15 tablets of placebo taken twice daily for 7 days and an additional 1 tablet for 1 day
Period: (PART A) Day 1, Day 3
Arm/Group | (PART A) Placebo Then Dalfampridine-ER 10mg | (PART A) Dalfampridine-ER 10mg Then Placebo | (PART B) Placebo Then Dalfampridine-ER 10mg | (PART B) Dalfampridine-ER 10mg Then Placebo
Started | 6 | 5 | 0 | 0
Completed | 6 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: (PART B) Day 1, Day 15
Arm/Group | (PART A) Placebo Then Dalfampridine-ER 10mg | (PART A) Dalfampridine-ER 10mg Then Placebo | (PART B) Placebo Then Dalfampridine-ER 10mg | (PART B) Dalfampridine-ER 10mg Then Placebo
Started | 0 | 0 | 12 | 12
Completed | 0 | 0 | 12 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population (Took at least one dose)
Groups:
- Total: Total of all reporting groups
Arm/Group | (PART A) Placebo Then Dalfampridine-ER 10mg | (PART A) Dalfampridine-ER 10mg Then Placebo | (PART B) Placebo Then Dalfampridine-ER 10mg | (PART B) Dalfampridine-ER 10mg Then Placebo | Total
Number analyzed (Participants) | 6 | 5 | 12 | 12 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (14.29) | 37.2 (9.39) | 41.1 (14.25) | 36.1 (14.04) | 37.05 (12.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 6 | 7 | 21
  Male | 2 | 1 | 6 | 5 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 3
  White | 3 | 4 | 11 | 10 | 28
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Dalfampridine-ER 10mg in Subjects With Cerebral Palsy (CP)
Description: Safety and tolerability will be assessed primarily by monitoring Treatment Emergent Adverse Events (TEAEs)
  TEAEs are defined as Adverse Events (AEs) with date of onset (or worsening) on or after the start-date of double-blind treatment and no more than 5 days after the last dose of double-blind treatment for Part A of the study and no more than 9 days for Part B of the study.
  The severity categories of mild, moderate or severe, are defined below:
  * Mild is defined as causing no limitation of usual activities
  * Moderate is defined as causing some limitation of usual activities
  * Severe is defined as causing inability to carry out usual activities
Time Frame: up to 31 days
Population: Safety Population (Took at least one dose)
Measure: Number; unit: participants
Groups:
- PART A: Placebo; PART A: Dalfampridine-ER 10mg: 6 subjects randomized into Sequence BA (placebo - dalfampridine-ER) 5 subjects randomized into Sequence AB (dalfampridine-ER - placebo)
  A single witnessed dose of placebo and a single witnessed dose of dalfampridine-ER 10 mg, two days apart
- PART B: Placebo; PART B: Dalfampridine-ER 10mg: 12 subjects randomized into Sequence BA (placebo - dalfampridine-ER) 12 subjects randomized into Sequence AB (dalfampridine-ER - placebo)
  Subjects received multiple doses of placebo and multiple doses of dalfampridine-ER 10mg
Arm/Group | PART A: Placebo | PART A: Dalfampridine-ER 10mg | PART B: Placebo | PART B: Dalfampridine-ER 10mg
Number analyzed (Participants) | 11 | 11 | 24 | 24
participants
  TEAEs | 1 | 2 | 6 | 9
  Serious TEAEs | 0 | 0 | 0 | 0
  TEAEs Maximum Severity - Mild | 1 | 2 | 5 | 8
  TEAEs Maximum Severity - Moderate | 0 | 0 | 1 | 1
  TEAEs Maximum Severity - Severe | 0 | 0 | 0 | 0
  TEAEs Possibly Related to Study Drug | 1 | 0 | 3 | 7
  TEAEs Leading to Withdrawal of Study Drug | 0 | 0 | 0 | 0

2. Secondary Outcome: Measure the Effects of Both Single and Multiple Doses of Dalfampridine-ER 10 mg on Sensorimotor Function
Description: * Hand strength as measured by a composite Z-score derived from the grip test, and key, tip and palmar pinch tests
  * Manual dexterity as measured by the Box and Block Test
  * Walking speed as measured by the Timed 25 Foot Walk (T25FW)
  * Gait as measured by gait analysis equipment (to be performed by sites that have the capability to perform it)
  * For Part B only, subjective impressions of treatment as measured by:
    * Subject Global Impression (SGI)
    * Clinician Global Impression (CGI)
Time Frame: up to 31 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 31 days
Description: Part A: up to 8 days Part B: up to 31 days
Arm/Group | PART A: Placebo | PART A: Dalfampridine-ER 10mg | PART B: Placebo | PART B: Dalfampridine-ER 10mg
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 1/11 | 2/11 | 6/24 | 9/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4.2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PART A: Placebo (N=11) | PART A: Dalfampridine-ER 10mg (N=11) | PART B: Placebo (N=24) | PART B: Dalfampridine-ER 10mg (N=24)
Headache (Nervous system disorders) | 0 | 2 | 1 | 3
Fatigue (General disorders) | 1 | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Joint crepitation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor (Acorda) has the right to review and comment on proposed publications within a specified time frame, up to 60 days; multi-center trials require joint publication unless specifically permitted otherwise.